CLINICAL TRIAL: NCT06708910
Title: Multiparametric 18F-FDG PET/MRI for Assessment and Prediction of Locoregional Therapy Response in HER2-positive Breast Cancer Patients Using Artificial Intelligence
Brief Title: AI-based pCR Assessment/Prediction in HER2-Positive BC Using PET/MRI
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University Hospital, Essen (Other); Marienhospital Bottrop (Unknown)
Responsible Party: Sponsor
Other Study IDs: 533909315; KI 2434/4-1 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: HER2 Positive Breast Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Weeks
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Goal of the observational study: Based on PET/MRI data it is possible to differentiate between complete and incomplete pathological remission after neoadjuvant systemic therapy in HER2-positive breast cancer patients.

The main question it aims to answer are:

Primary endpoint:

1) Sensitivity and specificity as co-primary endpoints for identification of HER2-positive breast carcinoma with complete pathologic remission (pCR; yT0 yN0) using 18F-FDG PET/MRI (response assessment)

Secondary endpoint(s):

1. Accuracy for the identification of patients with HER2-positive breast carcinoma with complete pathologic remission (pCR; yT0 yN0) using 18F-FDG PET/MRI (response assessment)
2. Sensitivity, specificity, and accuracy for the identification of patients with HER2-positive breast carcinoma with complete pathologic remission (pCR) of the primary (yT0) after neoadjuvant therapy using 18F-FDG PET/MRI (response assessment)
3. Sensitivity, specificity, and accuracy for the identification of patients with HER2-positive breast carcinoma with complete pathologic remission (pCR) of locoregional lymph node metastases (yN0) after neoadjuvant therapy using 18F-FDG PET/MRI (response assessment)
4. Evaluation of pre-treatment (baseline) 18F-FDG PET/MRI for predicting therapy response of the primary and locoregional lymph node metastases in patients with HER2-positive breast carcinoma supported by artificial-intelligence (prediction)
5. Evaluation of 18F-FDG PET/MRI for predicting therapy response of the primary in patients with HER2-positive breast carcinoma after the first cycles of systemic therapy supported by artificial-intelligence (prediction)
6. Evaluation of 18F-FDG PET/MRI for predicting therapy response of locoregional lymph node metastases in patients with HER2-positive breast carcinoma after the first cycles of system therapy supported by artificial-intelligence (prediction)

The guideline-recommended staging procedure (S3 Germany) using CT will be replaced by a whole-body 18F-FDG PET/MRI, including dedicated 18F-FDG PET/MRI of the breast. The histopathologic results of tissue samples obtained during routine clinical treatment after successful neoadjuvant systemic therapy will serve as a reference standard.

The study protocol involves the following examinations for all included patients:

1. Baseline (pre-treatment) examination to substitute for the staging examinations specified in the S3 guideline: Initial whole-body 18F-FDG PET/MRI including 18F-FDG PET/MRI of the breast
2. Thoracic 18F-FDG PET/MRI including 18F-FDG PET/MRI of the breast after the first two cycles of systemic therapy
3. Thoracic 18F-FDG PET/MRI including 18F-FDG PET/MRI of the breast after completion of systemic therapy and immediately before clinically indicated surgery

ELIGIBILITY:
Inclusion Criteria:

* Female
* HER2-positive breast carcinoma
* legally competent female patients aged ≥ 18 years
* willing and able to attend scheduled examinations
* written informed consent for study participation
* decision to receive neoadjuvant systemic therapy / exclusion of distant metastases

Exclusion Criteria:

* previous cancer diagnosis within the last five years or second, synchronous malignancy
* contraindication to MRI examination
* severe renal insufficiency
* pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In this study, we aim to enrol biological women with newly diagnosed HER2-positive breast carcinoma.
Study Population: In this study, we aim to enrol women with newly diagnosed HER2-positive breast carcinoma. For details please see Inclusion/Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Response assessment Primary EP | From enrollment to the end of treatment at 15 weeks
  Sensitivity and specificity as co-primary endpoints for identification of HER2-positive breast carcinoma with complete pathologic remission (pCR; yT0 yN0) using 18F-FDG PET/MRI

SECONDARY OUTCOMES:
Response assessment 1 | From enrollment to the end of treatment at 15 weeks
  Accuracy for the identification of patients with HER2-positive breast carcinoma with complete pathologic remission (pCR; yT0 yN0) using 18F-FDG PET/MRI
Response assessment 2 | From enrollment to the end of treatment at 15 weeks
  Sensitivity, specificity, and accuracy for the identification of patients with HER2-positive breast carcinoma with complete pathologic remission (pCR) of the primary (yT0) after neoadjuvant therapy using 18F-FDG PET/MRI
Response assessment 3 | From enrollment to the end of treatment at 15 weeks
  Sensitivity, specificity, and accuracy for the identification of patients with HER2-positive breast carcinoma with complete pathologic remission (pCR) of locoregional lymph node metastases (yN0) after neoadjuvant therapy using 18F-FDG PET/MRI
Prediction 1 | post baseline staging
  Evaluation of pre-treatment (baseline) 18F-FDG PET/MRI for predicting therapy response of the primary and locoregional lymph node metastases in patients with HER2-positive breast carcinoma supported by artificial-intelligence
Prediction 2 | 3 weeks post NAST start
  Evaluation of 18F-FDG PET/MRI for predicting therapy response of the primary in patients with HER2-positive breast carcinoma after the first cycles of systemic therapy supported by artificial-intelligence
Prediction 3 | 3 weeks post NAST start
  Evaluation of 18F-FDG PET/MRI for predicting therapy response of locoregional lymph node metastases in patients with HER2-positive breast carcinoma after the first cycles of system therapy supported by artificial-intelligence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Diagnostic and Interventional Radiology, Medical Faculty and University Hospital Duesseldorf, Heinrich-Heine-University Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No